CLINICAL TRIAL: NCT02007304
Title: Effects of Panax Ginseng and Salvia Miltiorrhiza Supplementation on Preventing Arterial Stiffening Effects Induced by Acute and Chronic Eccentric Exercise
Brief Title: Effects of Panax Ginseng and Salvia Miltiorrhiza Supplementation on Vascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201112068MIB
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Herbs (Experimental): participants assigned to experimental arm will take 300mg panax ginseng and 300mg salvia miltiorrhiza extracts in capsules for 12 weeks along with eccentric exercise training
  Interventions: Behavioral: Eccentric exercise training
- Placebo (Placebo Comparator): parcipants in this group will take placebo capsule containing microcrystalline cellulose
  Interventions: Behavioral: Eccentric exercise training

INTERVENTIONS:
Behavioral: Eccentric exercise training — 12 weeks of lower leg eccentric training

SUMMARY:
The purpose of is to determine the preventive effects of Chinese herb supplement with panax ginseng and salvia miltiorrhiza prior to eccentric resistance exercise on arterial stiffness and vascular reactivity by using a double-blind randomized control design and to examine the effects of a 12-week progressive eccentric resistance exercise training on arterial elasticity and vascular reactivity, and whether a long-term supplementation would ameliorate arterial stiffening effects elicited by exercise-induced inflammation and improve endothelial function.

ELIGIBILITY:
Inclusion Criteria:

-Healthy sedentary adults

Exclusion Criteria:

* obesity (BMI >30 kg/m2)
* smoking within past six months
* hypertension (high blood pressure >140/90 mmHg)
* personal history of diabetes (fasting blood glucose >126 mg/dL), heart disease, or other cardiovascular problems
* orthopedic injury that may prevent him or her from completing the exercise
* the use of over-the-counter supplements or vitamins

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Velocity | Before eccentric exercise and training
  PWV will be measured before, 6th week, 12th week of eccentric exercise training.
Pulse Wave Velocity | 6th week of eccentric exercise traininig
  PWV will be measured before, 6th week, 12th week of eccentric exercise training.
Pulse Wave Velocity | 12th week of eccentric exercise training
  PWV will be measured before, 6th week, 12th week of eccentric exercise training.

SECONDARY OUTCOMES:
Blood pressure | Before intervention
  Morning blood pressure will be measured before, during, and after 12 week of dietary and eccentric exercise intervention.
Blood pressure | 6th week of intervention
  Morning blood pressure will be measured before, 6th, and after 12 week of dietary and eccentric exercise intervention.
Blood pressure | 12th week of intervention
  Morning blood pressure will be measured before, during, and after 12 week of dietary and eccentric exercise intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Fu Lin, Ph.D, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Derived] Lin HF, Chou CC, Chao HH, Tanaka H. Panax ginseng and Salvia miltiorrhiza supplementation during eccentric resistance training in middle-aged and older adults: A double-blind randomized control trial. Complement Ther Med. 2016 Dec;29:158-163. doi: 10.1016/j.ctim.2016.10.003. Epub 2016 Oct 11. PMID 27912940
- [Derived] Lin HF, Tung K, Chou CC, Lin CC, Lin JG, Tanaka H. Panax ginseng and salvia miltiorrhiza supplementation abolishes eccentric exercise-induced vascular stiffening: a double-blind randomized control trial. BMC Complement Altern Med. 2016 Jun 6;16:168. doi: 10.1186/s12906-016-1139-4. PMID 27266702